CLINICAL TRIAL: NCT00211354
Title: Treatment of Retinal Vein Occlusion (RVO) With Open-Label Anecortave Acetate (15mg.)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Joan Daly,RN, LuEsther T. Mertz Retinal Research Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA in RVO
Expanded Access: Available
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — anecortave acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- anecortave acetate (Experimental): anecortave acetate 15 mg. juxtascleral injection every 6 months for 24 months
  Interventions: Drug: Anecortave Acetate

INTERVENTIONS:
Drug: Anecortave Acetate — ancortave acetate 15 mg. juxtascleral injection every 6 months for 24 months.
  Other Names: retaane

SUMMARY:
Retinal Vein Occlusion is a blockage of the blood vessels that drain out of the retina. Complications of retinal vein occlusion which threaten vision include neovascularization(growth of new blood vessels)and macular edema ( accumulation of fluid "leaking" from abnormal blood vessels). Currently, the treatment of retinal vein occlusion is laser photocoagulation. This treatment has found to have limited use in this type of condition.Anecortave Acetate is being considered as an attempt to control the growth of the abnormal blood vessels.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of patients Retinal Vein Occlusion.
2. Patients must be 18 years of age or older to receive treatment.
3. Visual acuity of 20/30 to 20/320 Study Eye on the ETDRS visual acuity chart.
4. Visual acuity of 20/800 or better Fellow Eye on the ETDRS visual acuity chart.

Exclusion Criteria:

1. Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
2. Patients who have undergone intraocular surgery within last 2 months.
3. Patient participating in any other investigational drug study.
4. Use of an investigational drug or treatment related or unrelated to their condition within 30 days prior to receipt of study medication.
5. Inability to obtain photographs to document CNV (including difficulty with venous access).
6. Patient with significant liver disease or uremia.
7. Patient with known adverse reaction to fluorescein and indocyanine green or iodine.
8. Patient has a history of any medical condition which would preclude scheduled visits or completion of study.
9. Patient has had insertion of scleral buckle in the study eye.
10. Patient has received radiation treatment.
11. Patient is on anticoagulant therapy with the exception of aspirin.
12. Patient is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-03; Primary Completion 2007-03 (Estimated); Study Completion 2007-04 (Estimated)

PRIMARY OUTCOMES:
to investigate the use of anecortave acetate for treatment of retinal vein occlusion | 24 months

SECONDARY OUTCOMES:
mean change of VA (ETDRS) from baseline to 24 months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A. Yannuzzi, MD, Principal Investigator — Manhattan Eye, Ear & Throat Hospital
Locations (1):
- Manhattan Eye, Ear & Throat Hospital, New York, New York, United States